CLINICAL TRIAL: NCT03081078
Title: Effects of Community-based Caring Contact on Post-discharge Young Adults With Self-harm - a Multi-center Randomized Controlled Trial
Brief Title: Effects of Community-based Caring Contact on Post-discharge Young Adults With Self-harm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); United Christian Hospital (Other); North District Hospital (Other); Pamela Youde Nethersole Eastern Hospital (Other)
Responsible Party: Principal Investigator, Dr.Yik-Wa Law, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HKU-ECS-27612816
Record Dates: First submitted 2017-03-03; First posted 2017-03-15 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Self Inflicted Injury; Suicide and Self Inflicted Injury
MeSH Terms: conditions — Self-Injurious Behavior; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TAU w/ mobile app + volunteer support (Experimental): Participants will be receiving usual medical treatment from the hospitals with a mobile app engagement intervention, plus support from volunteers.
  Interventions: Behavioral: Volunteer support; Other: Mobile app
- TAU w/ mobile app engagement (Experimental): Participants will be receiving usual medical treatment from the hospitals with a mobile app engagement intervention.
  Interventions: Other: Mobile app
- Treatment as Usual (TAU) (No Intervention): Participants will be receiving usual medical treatment from the hospitals, and without the interventions (i.e., mobile app and/or volunteer support) introduced through this randomized control trial.

INTERVENTIONS:
Behavioral: Volunteer support — Each participant will be matched with a pair of trained volunteers (under pre-determined safety measures), who will initiate caring contact via telephone or text messages at least twice a month for two months. Participants will be free to respond or not.
  Arms: TAU w/ mobile app + volunteer support
Other: Mobile app — Participants will receive programmed care messages and reminders of community resources and healthcare contacts on a regular basis. The app will also provide simple self-help mood checking and relaxation exercises.
  Other Names: Mobile app engagement
  Arms: TAU w/ mobile app + volunteer support; TAU w/ mobile app engagement

SUMMARY:
The study will determine whether community-based caring contact via a mobile app connection with or without volunteer support in addition to treatment as usual (psychiatric and psychosocial treatments) has an effect on suicidal ideation and treatment compliance among post-discharge self-harm young adults.

DETAILED DESCRIPTION:
The proposed study will determine whether community-based caring contact via a mobile app connection with or without volunteer support in addition to treatment as usual (TAU; psychiatric and psychosocial treatments) is effective in reducing suicidal ideation, enhancing treatment compliance, reducing thwarted belongingness and perceived burdensomeness and hopelessness among post-discharge self-harm young adults, and if personalized contact by volunteers has additional effects reducing suicidal ideation among post-discharge self-harm individuals.

108 participants aged 18-45 with an index self-harm episode will be recruited from the Accident & Emergency Department (AED) of 4 local public hospitals, and randomized into the TAU, mobile app group with, and without volunteer support. Each participant will complete a questionnaire at the 4 measurement time points at baseline (T0), one-month (T1) and the end of the 2-month intervention period (T2), and post-intervention at the three-month point (T3) from the baseline. The primary outcomes include Suicidal ideation, hopelessness, thwarted belongingness & perceived burdensomeness, treatment (TAU) compliance, and suicidality.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with an index episode of self-poisoning or self-injury with or without suicide intent, based on the ICD-10 codes for self-harm with and without suicide intent (i.e., X60 to X84 and R45.8)
* Admission to the AEDs at the 4 collaborating public hospitals in Hong Kong (United Christian Hospital, North District Hospital, Queen Mary Hospital, and Pamela Youde Nethersole Eastern Hospital)
* Mentally well assessed by a psychiatrist or Consultation Liaison Nurses (CLNs)
* Capable of providing written Informed Consent Form

Exclusion Criteria:

* Individuals with DSM-IV-TR Axis II disorder; or
* Individuals with severe psychotic mental illness or bipolar disorder

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Adult Suicidal Ideation at 1-month, 2-month and 3-month | Baseline, 1 month, 2 months, 3 months
  Change in scores on Suicidal ideation as measured by the self-report the Adult Suicidal Ideation Questionnaire - the four-item short form in Chinese (ASIQ-4) (Fu, Liu, & Yip, 2007)
Change from baseline Measurement of Hopelessness at 1-month, 2-month and 3-month | Baseline, 1 month, 2 months, 3 months
  Change in scores on Hopelessness as measured by a self-report 4-item short-form of Beck Hopelessness Scale Chinese version (BHS-4) (Beck, Weissman, Lester, & Trexler, 1974; Yip & Cheung, 2006; Shek, 1993).
Change from baseline Interpersonal Needs at 1-month, 2-month and 3-month | Baseline, 1 month, 2 months, 3 months
  Change in scores on Thwarted Belongingness (TB) and Perceived Burdensomeness (PB) as measured by the Interpersonal Needs Questionnaire (INQ-15), a 15-item measure of beliefs about whether one's need to belong is met or unmet and self-perceptions of being a burden to others (Van Orden, 2012).
Change from baseline Service Utilization at 1-month, 2-month and 3-month | Baseline, 1 month, 2 months, 3 months
  Self-reported compliance with prescribed treatment (frequency) in relation to the index self-harm episode, including psychiatric follow-up care (e.g., medication, out-patient follow-up treatment, and community psychiatric nursing service) and psycho-social services (e.g., clinical psychology service, medical social work service, etc.) as measured by a self-developed service utilization checklist.
Change from baseline Suicidality at 1-month, 2-month and 3-month | Baseline, 1 month, 2 months, 3 months
  Suicidality as measured by a four-item scale for levels of suicidality in the past 12 months (Centre for Suicide Research and Prevention, The University of Hong Kong, 2005)

SECONDARY OUTCOMES:
Change from baseline Depressive state at 1-month, 2-month and 3-month | Baseline, 1 month, 2 months, 3 months
  Depressive state as measured by the Center for Epidemiologic Studies Depression Scale (CES-D) (Lam et al., 2004).
Change from baseline Self-harming repetition at 1-month, 2-month and 3-month | Baseline, 1 month, 2 months, 3 months
  Self-reported frequency of self-harm repetition (retrieved from the Hong Kong Special Administrative Region (HKSAR) Coroner's Court)
Change from baseline suicide deaths at 1-month, 2-month and 3-month | Baseline, 1 month, 2 months, 3 months
  Number of suicide deaths (retrieved from the Hong Kong Special Administrative Region (HKSAR) Coroner's Court)
Change of baseline index self-harm episode | Baseline, 1 month, 2 months, 3 months
  Hospital records on the details of index self-harm episode including clinical diagnosis, treatment received, discharged information and number of Accident & Emergency Department (AED) re-admissions, etc. in Clinical Management System (CMS), Outpatient Appointment System (OPAS), and Accident & Emergency Department Clinical Information System (AEIS)
Demographic and socioeconomic information | Baseline
  Questionnaire on participants' demographic and socioeconomic information (e.g. Sex, Date of birth, birth place, years living in Hong Kong, Marital status, religion, residential district, education, living status, employment, occupation, social security, etc.
Change of time spent on each programme activity of the app at 1-months, 2-months | From Baseline to 2 months
  The log-in time-stamp of each activity (including but not limited to reviewing the information or messages provided on the app, pattern of using the app, etc.)
Change of time spent and type of contact made by volunteers with participants at 1-months, 2-months | 1-month, 2-months
  Volunteer service records on time-stamp of each type of contact (i.e. in-person, phone contact, letters & email, and social media)
Final and Monthly Qualitative Description on participants' progress | up to 3 months
  Reported by volunteers. items included case summary, services offered, volunteer-participant relationship, follow-up plan, self-reflection and areas of improvement, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Yik-wa Law, PhD, Principal Investigator — The University of Hong Kong
Locations (4):
- Hong Kong (4):
  - Pamele Youde Nethersole Eastern Hospital, Chai Wan, Eastern District
  - United Christian Hospital, Sau Mau Ping, Kwun Tong District
  - North District Hospital, Sheung Shui, North District
  - Queen Mary Hospital, Central, Southern District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Law YW, Yip PS, Lai CC, Kwok CL, Wong PW, Liu KS, Ng PW, Liao CW, Wong TW. A Pilot Study on the Efficacy of Volunteer Mentorship for Young Adults With Self-Harm Behaviors Using a Quasi-Experimental Design. Crisis. 2016 Nov;37(6):415-426. doi: 10.1027/0227-5910/a000393. Epub 2016 Jun 9. PMID 27278570
- [Background] Luxton DD, June JD, Comtois KA. Can postdischarge follow-up contacts prevent suicide and suicidal behavior? A review of the evidence. Crisis. 2013 Jan 1;34(1):32-41. doi: 10.1027/0227-5910/a000158. PMID 22846445
- [Background] Van Orden KA, Cukrowicz KC, Witte TK, Joiner TE. Thwarted belongingness and perceived burdensomeness: construct validity and psychometric properties of the Interpersonal Needs Questionnaire. Psychol Assess. 2012 Mar;24(1):197-215. doi: 10.1037/a0025358. Epub 2011 Sep 19. PMID 21928908
- [Derived] Law YW, Lok RHT, Chiang B, Lai CCS, Tsui SHM, Chung PYJ, Leung SC. Effects of Community-Based Caring Contact in Reducing Thwarted Belongingness Among Postdischarge Young Adults With Self-Harm: Randomized Controlled Trial. JMIR Form Res. 2023 Aug 16;7:e43526. doi: 10.2196/43526. PMID 37585260
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617